CLINICAL TRIAL: NCT00888563
Title: Fatigue in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090131; 09-NR-0131
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-11-16

CONDITIONS: Healthy Volunteer; Fatigue; Depression
Keywords: Fatigue; Depression; Healthy Volunteer; HV
MeSH Terms: conditions — Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* People with many different diseases have symptoms of fatigue, which is a general sense of tiredness; however, the causes are not fully understood. Fatigue symptoms may be related to a person s level of fitness, health, and blood chemistries.
* Researchers are studying the potential role of plasma cytokines (signaling molecules) and hypothalamic-pituitary-adrenal (HPA) axis (part of the neuroendocrine system that controls stress) functioning in symptoms of fatigue.

Objectives:

* To characterize the symptoms of fatigue in healthy individuals.
* To collect information on fatigue, pain, depression, stress, sleepiness, and quality of life from healthy adults of all ages.
* To compare results obtained from people with various illnesses to better understand possible causes of fatigue that are associated with those diseases.

Eligibility:

* Physically and mentally healthy volunteers18 years of age or older who can speak and read the English language.
* Exclusion criteria include individuals with a disease or condition causing significant fatigue (congestive heart failure, cancer, or sleep disorders), individuals taking medicines that cause fatigue (beta blockers, diuretics, or narcotics), and individuals who have a major psychiatric condition (major depression, anxiety disorder, or schizophrenia).
* The following individuals may not participate: those who have two more alcoholic drinks per day, who use illicit drugs, or who drink more than 4 cups of coffee, 8 cups of soda or tea, or similar amounts of other caffeine-containing beverages a day, or eat more than 1 pound of chocolate per day; and individuals who worked evenings or night shifts in the past month.
* Women who are pregnant or breastfeeding are not eligible.

Design:

* Participants must make two outpatient visits to the Clinical Center. Each visit will last 5 hours and participants must refrain from smoking and consuming alcohol and caffeine for at least 24 hours.
* During the first study visit, researchers will conduct the following tests:

  * Psychiatric interview, medical history, pregnancy test, and drug test.
  * Urine test to measure the levels of stress hormones.
  * Questionnaires that measure fatigue, pain, depression, stress, daytime sleepiness, and activity.
  * Physical fitness test, including strength tests, walking tests, and physical activity monitoring.
* Before the second study visit, patients must refrain from smoking and consuming caffeine and alcohol for at least 24 hours and have nothing, even water, by mouth after midnight. During the second study visit, the following tests will be conducted:

  * Stress hormone test (participant will receive a cortisol-releasing hormone).
  * Four intravenous blood draws to determine cytokine profiles, gene expression, and levels of stress hormones (immune and gentic analysis).
* Participants will receive a small financial compensation for participation in the study.

DETAILED DESCRIPTION:
This protocol is designed to characterize the symptoms of fatigue in healthy individuals using standardized questionnaires and determine if physical activity, pain, depression, fatigue

catastrophizing, stress, and daytime sleepiness play a role in the experience. This study will also examine the potential role of plasma cytokines and hypothalamic-pituitary-adrenal axis (HPA) functioning in symptoms of fatigue in healthy individuals.

Eligible participants will complete questionnaires that measure fatigue, pain, depression, fatigue catastrophizing, perceived stress, daytime sleepiness, neurological health, and physical activity. Participants will also perform strength testing (e.g. hand grips), walk testing (6-minute walk test), exercise testing on a treadmill, and physical activity monitoring using a portable activity device. Blood samples will be obtained to determine cytokine profiles, gene expression, and levels of stress hormones (cortisol, dehydroepiandrosterone [DHEA], catecholamines). Urine samples will also be obtained to measure the levels of stress hormones excreted. Information collected in this protocol will be used to make comparison in subjects who experience extreme symptoms of fatigue due to many different disorders, in order to better understand the mechanisms of fatigue.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, participants must meet the following:

* Healthy, 18 years of age or older;
* Speak and understand the English language.

EXCLUSION CRITERIA:

Participants with any one of the following will be excluded:

* Inability to provide informed consent for the study;
* Are unwilling or unable to cooperate with the study procedures or travel to NIH for the procedures;
* Have a confirmed medical condition causing clinically significant fatigue symptom (e.g. congestive heart failure, cancer actively receiving therapy, sleep disorders);
* Currently taking medications that cause fatigue (e.g. diuretics, beta blockers, narcotics);
* Working late evening and night shifts within the past month;
* Have severe psychiatric conditions (e.g. major depressive disorder, bipolar disorder, anxiety disorder, schizophrenia, drug and/or addiction abuse or dependence);
* Report consuming more than 300mg of caffeine containing beverages (approximately 4 cups of coffee or 8 cups of soda or tea) or food (approximately 1 lb of chocolate) within 24 hours;
* Reports consuming more than 2 servings of alcohol containing beverages every day and with detectable blood alcohol content (BAC) using breath analyzer (greater than 1 mg/dL of BAC);
* Pregnant or lactating women.
* Unable to refrain from smoking at least 4 hours prior to exercise testing sessions
* Any medical condition that limits exercise performance (e.g. any condition with a ventilatory limitation during maximal exercise)
* Any medical condition that affects participants safety with exercise (e.g.: severe heart disease, uncontrolled diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-04-23; Study Completion 2017-11-16

PRIMARY OUTCOMES:
fatigue score of healthy individuals using standardized questionnaires. | study completed

SECONDARY OUTCOMES:
Physical activity, pain, depression, stress, and daytime sleepiness scores; the HPA axis function of healthy individuals; the proinflammatory cytokine profile and gene expression in response to stress. | study completed

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Levy M. Cancer fatigue: a review for psychiatrists. Gen Hosp Psychiatry. 2008 May-Jun;30(3):233-44. doi: 10.1016/j.genhosppsych.2008.01.004. PMID 18433655
- [Background] Krupp LB, Pollina DA. Mechanisms and management of fatigue in progressive neurological disorders. Curr Opin Neurol. 1996 Dec;9(6):456-60. doi: 10.1097/00019052-199612000-00011. PMID 9007405
- [Background] Brola W, Ziomek M, Czernicki J. [Fatigue syndrome in chronic neurological disorders]. Neurol Neurochir Pol. 2007 Jul-Aug;41(4):340-9. Polish. PMID 17874343
- [Derived] Flynn S, Leete J, Shahim P, Pattinson C, Guedes VA, Lai C, Devoto C, Qu BX, Greer K, Moore B, van der Merwe A, Ekanayake V, Gill J, Chan L. Extracellular vesicle concentrations of glial fibrillary acidic protein and neurofilament light measured 1 year after traumatic brain injury. Sci Rep. 2021 Feb 16;11(1):3896. doi: 10.1038/s41598-021-82875-0. PMID 33594224
- [Derived] Lukkahatai N, Walitt B, Espina A, Gelio A, Saligan LN. Understanding the Association of Fatigue With Other Symptoms of Fibromyalgia: Development of a Cluster Model. Arthritis Care Res (Hoboken). 2016 Jan;68(1):99-107. doi: 10.1002/acr.22626. PMID 26017904